CLINICAL TRIAL: NCT03124485
Title: Prospective Randomized Trial Comparing Endoscopic Sleeve Gastroplasty Versus Conventional Laparoscopic Sleeve Gastrectomy in Patients With Morbid Obesity: From Physical and Functional Outcomes to Changes in Hormonal Profiles
Brief Title: Endoscopic Sleeve Gastroplasty for Morbid Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Enders K.W. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRE2017.127-T
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Endoscopic Sleeve Gastroplasty

STUDY DESIGN:
Intervention Model Description: This study protocol aims to test the hypothesis that endoscopic sleeve gastroplasty (ESG) IS NOT inferior to conventional laparoscopic surgical sleeve gastrectomy (LSG) in terms of weight loss and improvement of glycemic control for Asian obese patients. It also investigates and compares the safety profile, improvement of co-morbidities, functional outcomes and changes in gut hormone profiles between the two bariatric procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Sleeve Gastroplasty (Experimental): A series of full thickness sutures done with Overstitch in the triangular stitch pattern as mentioned by Lopez-Nava[29] will be placed according to the APC markings. The suturing is initiated from the antrum distally and moved proximally towards the gastric fundus. A total of 6 to 8 plications are placed to reduce the gastric lumen. Five sham dressings would also be applied to patient's abdominal wall during the first week to minimize the bias in pain scoring.
  Interventions: Procedure: Endoscopic Sleeve Gastroplasty
- Laparoscopic Sleeve Gastrectomy (Active Comparator): Sleeve gastrectomy is then performed using lapaorscopic linear staplers, starting from a point 5-6cm proximal to the pylorus up to the angle of His along the left side of the Mid-sleeve tube. Haemostasis of the staple line is secured by suture plication with the Mid-sleeve tube in situ to ensure no compromise of the gastric tube lumen. All the wounds are closed with staples after local anaesthetic infiltration and covered with non-transparent dressings.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Endoscopic Sleeve Gastroplasty — An oesophageal overtube is then inserted to facilitate passage of the endoscope mounted with Overstitch device. A series of full thickness sutures done with Overstitch in the triangular stitch pattern as mentioned by Lopez-Nava[29] will be placed according to the APC markings. The suturing is initiated from the antrum distally and moved proximally towards the gastric fundus. A total of 6 to 8 plications are placed to reduce the gastric lumen. Five sham dressings would also be applied to patient's abdominal wall during the first week to minimize the bias in pain scoring.
  Arms: Endoscopic Sleeve Gastroplasty
Procedure: Laparoscopic Sleeve Gastrectomy — Sleeve gastrectomy is then performed using lapaorscopic linear staplers, starting from a point 5-6cm proximal to the pylorus up to the angle of His along the left side of the Mid-sleeve tube. Haemostasis of the staple line is secured by suture plication with the Mid-sleeve tube in situ to ensure no compromise of the gastric tube lumen. All the wounds are closed with staples after local anaesthetic infiltration and covered with non-transparent dressings.
  Arms: Laparoscopic Sleeve Gastrectomy

SUMMARY:
Obesity and its related metabolic disorders are increasingly a heavy health burden to many parts of the world. Weight control is a well-known important step in avoiding type 2 diabetes mellitus (T2DM). It is also an essential component for normalizing the blood glucose and preventing macrovascular and microvascular insults to patients with diagnosed T2DM. However, life-style modification, physical exercise and dietary adjustment are ineffective measures which are unlikely to confer adequate and sustainable weight loss for the truly obese. On the other hand, large scale long-term follow-up studies have confirmed the role of bariatric surgery in providing durable weight loss and remarkable improvement on medical comorbidities. Among all the bariatric operations, laparoscopic sleeve gastrectomy (LSG) is currently the most widely adopted procedure worldwide because of its simplicity and effectiveness in weight reduction. However, LSG is not without risk. Staple-line hemorrhage, leakage and stenosis are potentially life-threatening complications. LSG is also costly because of the need for expensive laparoscopic staplers.

DETAILED DESCRIPTION:
A new endoscopic bariatric therapy, namely endoscopic sleeve gastroplasty (ESG), has recently been proposed as a non-surgical procedure for the management of obesity with or without diabetes mellitus. Preliminary data based on single arm series or phase II studies have reported promising short and intermediate term weight control effect.

However, whether ESG is a feasible option comparable to LSG in the intermediate term remains an unanswered question. In addition, physical and functional outcomes after ESG were not well documented in most of the reported series.

Realizing there is a knowledge gap in applying ESG to patients with morbid obesity, we propose to study and compare the efficacy of weight control and functional outcomes of ESG against conventional LSG. Through this prospective randomized trial, the safety profiles, quality of life and changes in fasting and post-prandial gut hormone secretion after the two procedures will also be assessed and compared. The evidence thus generated shall lay a scientific foundation for ESG which may become an alternative choice for patients who have concerns about complication and irreversibility of most bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A BMI > 35 kg/m2
2. A BMI > 30 kg/m2 with T2DM
3. A BMI>3 30kg/m2 with 2 or more co-morbidities

Exclusion Criteria:

1. Significant anaesthetic risk (> ASA III)
2. History of diabetic ketoacidosis or hyperosmolar coma
3. Uncontrolled T2 DM with HbA1c > 12%
4. A BMI > 45 kg/m2
5. Malignancy diagnosed within 5 years
6. Endoscopic findings of any pre-neoplastic/neoplastic lesions, portal hypertensive gastropathy or significant varices
7. Chronic renal failure requiring dialysis
8. Previous upper abdominal surgery (including bariatric surgery) affecting gastroduodenal configuration
9. Major psychiatric illness including major depression and substance abuse
10. Pregnancy or ongoing breast-feeding
11. Inmates

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of excess weight loss | 1 year

SECONDARY OUTCOMES:
operative time | during operation
total blood loss intra-operation | during operation
  total blood loss will be recorded in operation record
early postoperative pain scores | 7 days
perioperative complications | 30 days
  mortality
postoperative hospital stay | 30 days
Percentages of excess weight loss | 1 year
  (%EWL)
total weight loss | 1 year
  (%TWL)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided